CLINICAL TRIAL: NCT01819623
Title: Effect of Non-pharmacological Therapy on Cognitive Function of Patients With Cognitive Impairment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Financial issues (no participants enrolled)
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, José Alberto Ávila Funes, MD, PhD, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GER-830-13/14-1
Record Dates: First submitted 2013-03-11; First posted 2013-03-27 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Cognitive training
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-pharmacological therapy (Experimental): This group will be supervised nonpharmacologic therapy
  Interventions: Other: Non-pharmacological therapy
- Control (No Intervention): This group will receive the standard treatment for mild cognitive impairment

INTERVENTIONS:
Other: Non-pharmacological therapy — It consists of a weekly two-hour session. During the first hour yoga classes will taught by teacher, during second hour supervised cognitive training by a psychologist based on Memory Program designed by Memory Unit of Madrid
  Other Names: Supervised nonpharmacologic therapy
  Arms: Non-pharmacological therapy

SUMMARY:
Supervised nonpharmacologic therapy improve cognitive function in patients with Mild Cognitive Impairment

ELIGIBILITY:
Inclusion Criteria:

* Patients 60 years and older with Mild Cognitive Impairment according to Petersen Criteria
* Phone number available

Exclusion Criteria:

* Untreated depression
* Evidence of a reversible cause of cognitive decline
* Dementia of any type and stage
* Severe sensory deficit unresolved
* Metastatic cancer
* Hemoglobin level < 8g/dL
* Chronic Obstructive Pulmonary Disease Gold stage 3 or 4
* Congestive Heart Failure decompensated, unstable angina o Functional Class IV according to New York Heart Association
* Participation in another protocol that prevents its participation in this research
* Chronic use of benzodiazepines, tricyclic antidepressants
* Patients whose place of residence can not attend the sessions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | six months
  Cognitive function measured by Alzheimer's Disease Assessment Cognitive Scale (ADAS-Cog) sum of boxes after non-pharmacological intervention for six months.

SECONDARY OUTCOMES:
Cognitive function six months after completing intervention | one year
  Cognitive function measured by Alzheimer's Disease Assessment Cognitive Scale (ADAS-Cog) six months after completing intervention
Depressive symptoms | six months
  Depressive symptoms measured by Geriatric Depression Scale (GDS) before and after intervention period

OTHER OUTCOMES:
quality of life | six months
  Quality of life measured by a scale validated in Spanish before and after intervention period

CONTACTS AND LOCATIONS:
Overall Officials: JOSÉ ALBERTO MD ÁVILA, Geriatrician, Principal Investigator — National Institute of Medical Sciences and Nutrition Salvador Zubirán
Locations (1):
- National Institue of Medical Sciences and Nutrition Salvador Zubirán, Mexico City, Mexico City, Mexico